CLINICAL TRIAL: NCT03504410
Title: Phase 3 Multicenter Randomized Trial to Evaluate Efficacy and Safety of CPI-613 in Combination With HD Cyt. and Mito. vs HD Cyt. and Mito. Therapy and Control Sub-groups in Older Patients With R/R AML
Brief Title: Efficacy/Safety of CPI-613 in Combination With HD Cyt. and Mito. vs HD Cyt. and Mito. in Older Patients With R/R AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futile
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML003
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Results first posted 2022-12-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — devimistat; Cytarabine; Mitoxantrone; Etoposide; fludarabine; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPI-613 + HD Cytarabine and Mitoxantrone (Experimental): CPI-613 + High Dose Cytarabine and Mitoxantrone
  CPI-613 at 2,000 mg/m2/day from day 1 to 5.
  Cytarabine at 1gm/m2 (5 doses), every 12 hours starting day 3. Mitoxantrone at 6gm/m2 (3 doses), everyday following the 1st, 2nd and 5th doses of Cytarabine.
  Interventions: Drug: CPI-613 + High Dose Cytarabine and Mitoxantrone
- Control (HAM) and control sub-groups (MEC and FLAG) (Active Comparator): High Dose Cytarabine and Mitoxantrone
  Cytarabine at 1gm/m2 (5 doses), every 12 hours starting day 3. Mitoxantrone at 6gm/m2 (3 doses), everyday following the 1st, 3rd and 5th doses of Cytarabine.
  Mitoxantrone, Etoposide and Cytarabine
  Etoposide 80mg/m over 60 minutes as a central line IV infusion; 6 doses Day 1 though 6 Cytarabine 1000mg/m2 over 3 hours as a central line IV infusion: 6 doses, Day 1 through 6 Mitoxantrone 6 mg/m2 over 30 minutes as a central line IV infusion: 6 dose, Day 1 through 6
  Fludarabine, Cytarabine and Filgrastim
  Fludarabine 30mg/m2/day over 30 minutes as a central line IV infusion; 5 doses Day 1 though 5 Cytarabine 2g/m2 over 4 hours as a central line IV infusion: 4 hours after Fludarabine: 5 doses, Day 1 through 5 Filgrastim 5µg/kg/day by SQ or as per institutional guidelines starting from Day 1 through Day 5
  Interventions: Drug: High Dose Cytarabine and Mitoxantrone; Drug: Mitoxantrone, Etoposide and Cytarabine; Drug: Fludarabine, Cytarabine, Filgrastim

INTERVENTIONS:
Drug: CPI-613 + High Dose Cytarabine and Mitoxantrone — CPI-613 + High Dose Cytarabine and Mitoxantrone CPI-613: 2000mg/m2, 5 doses once a day, days 1-5 Cytarabine 1gm/m2, 5 doses every 12hrs starting day 3 through day 5 Mitoxantrone 6mg/m2, 3 doses, once a day following the first, third and fifth doses of Cytarabine
  Other Names: CPI-613, CHAM
  Arms: CPI-613 + HD Cytarabine and Mitoxantrone
Drug: High Dose Cytarabine and Mitoxantrone — Cytarabine 1gm/m2, 5 doses every 12hrs starting day 3 through day 5 Mitoxantrone 6mg/m2, 3 doses, once a day following the first, third and fifth doses of Cytarabine
  Other Names: HAM
  Arms: Control (HAM) and control sub-groups (MEC and FLAG)
Drug: Mitoxantrone, Etoposide and Cytarabine — Mitoxantrone, Etoposide and Cytarabine
  Etoposide 80mg/m over 60 minutes as a central line IV infusion; 6 doses Day 1 though 6 Cytarabine 1000mg/m2 over 3 hours as a central line IV infusion: 6 doses, Day 1 through 6 Mitoxantrone 6 mg/m2 over 30 minutes as a central line IV infusion: 6 dose, Day 1 through 6
  Other Names: MEC
  Arms: Control (HAM) and control sub-groups (MEC and FLAG)
Drug: Fludarabine, Cytarabine, Filgrastim — Fludarabine, Cytarabine and Filgrastim
  Fludarabine 30mg/m2/day over 30 minutes as a central line IV infusion; 5 doses Day 1 though 5 Cytarabine 2g/m2 over 4 hours as a central line IV infusion: 4 hours after Fludarabine: 5 doses, Day 1 through 5 Filgrastim 5µg/kg/day by SQ or as per institutional guidelines starting from Day 1 through Day 5
  Other Names: FLAG
  Arms: Control (HAM) and control sub-groups (MEC and FLAG)

SUMMARY:
A Phase III study to evaluate the safety and efficacy of CPI-613® (devimistat) in combination with High Dose Cytarabine and Mitoxantrone in comparison with high dose Cytarabine and Mitoxantrone and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in older patients with relapsed/refractory Acute Myeloid Leukemia. CPI-613® (devimistat) targets the altered energy metabolism and processes for production of ATP and essential bio-intermediates unique to and characteristic of most cancer cell types. The addition of CPI-613® (devimistat) to high dose cytarabine and mitoxantrone (CHAM) will improve the complete remission (CR) rate in patients 50 years or older with relapsed or refractory AML when compared to HAM alone or other control sub groups.

DETAILED DESCRIPTION:
Subjects were randomized in 1:1 allocation ratio by IWRS according to the stratification factors. However, the control sub-groups (MEC and FLAG) were capped at 100 (50 per sub-group).

Subjects in both Arm 1 and Arm 2 were planned to receive induction cycle 1 treatment for at least 14 days. Subjects will receive follow-up therapy based on results of the bone marrow aspirate, and CR/complete remission with incomplete recovery (CRi) status.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient has provided an informed consent prior to initiation of any study specific activities/procedures
2. Males and females age ≥ 50 years must have histologically documented AML that is relapsed from, or refractory to, prior standard therapies
3. Refractory is defined as failure to achieve CR or CRi following:

   1. At least one cycle of any anthracycline, cytarabine or fludarabine containing induction regimen or persistence of disease on a nadir marrow following at least one cycle of any anthracycline, cytarabine or fludarabine containing induction regimen
   2. Persistent disease after at least 2 cycles of a hypomethylating agent (azacytidine or decitabine) with or without venetoclax
4. Relapse is defined as development of recurrent AML (as described by Döhner et al, 2017)6 after CR or CRi has been achieved with a prior chemotherapy or after disease progression on a hypomethylating agent with or without venetoclax
5. ECOG PS 0-2
6. Expected survival greater than 3 months
7. Women of child-bearing potential (i.e. women who are pre-menopausal or < 2 years post menopausal or not surgically sterile) must practice a highly effective method of birth control consistent with local regulations regarding the use of birth control methods. Examples: use of oral, injected or implanted hormonal methods of contraception; placement of an intra uterine device (IUD) or intrauterine system (IUS); male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence during and for 6 months after the last administered dose of CHAM or HAM therapy and control sub-groups (MEC and FLAG), and must have a negative serum pregnancy test within 1 week prior to treatment initiation and at 1st day of each cycle and at the end of systemic exposure. (Note: pregnant patients are excluded because the effects of CPI-613® (devimistat) on a fetus are unknown)
8. Fertile men who are sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository during the study period and up to 6 months after completion of the study screening, unless documentation of infertility exists
9. Good state of mental health, ability to understand and willingness to sign the informed consent form (ICF)
10. No radiotherapy, treatment with cytotoxic chemotherapy, treatment with biologic agents or any anti-cancer therapy for R/R AML within the 1 week prior to treatment with CPI-613® (devimistat). Hydroxyurea and/or venetoclax and oral tyrosine kinase (FLT3) or Isocitrate Dehydrogenase 1 and 2 (IDH1/2), BCL-2 or hedgehog inhibitors being used with Grade ≤ 2 toxicity can be taken until the day prior to starting of CHAM or HAM therapy or control sub-groups (MEC and FLAG). Previous exposure to a hypomethylating agent either alone or in combination with Isocitrate Dehydrogenase 1 and 2 (IDH1/2), BCL-2 or hedgehog inhibitors are allowed until the day prior to starting of CHAM or HAM therapy and control sub-groups (MEC and FLAG). Patients must have fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities with the exception of alopecia (returned to baseline status as noted before most recent treatment). Patients with persisting, non-hematologic, non-infectious toxicities from prior treatment Grade ≤ 2 are eligible but must be documented as such
11. Laboratory values ≤ 2 weeks before dosing must be:

    * Adequate hepatic function (aspartate aminotransferase/serum glutamic-oxaloacetic transaminase [AST/SGOT] ≤ 5 x upper limit of normal [ULN], alanine aminotransferase/serum glutamic oxaloacetic transaminase [ALT/SGPT] ≤ 5 × ULN, bilirubin ≤ 1.5 × ULN)
    * Adequate renal function (serum creatinine clearance ≥ 60 mL/min per CockCroft Gault formula)
    * Adequate coagulation (International Normalized Ratio [INR] must be < 1.7 unless on vitamin k antagonist anticoagulation)
12. Left Ventricular Ejection Fraction (LVEF) by Transthoracic Echocardiogram (TTE) or Multigated Acquisition Scan (MUGA) or cardiac Magnetic Resonance Imaging (MRI), sufficient to safely administer mitoxantrone. Subjects must have an LVEF ≥ 45%
13. No marked baseline prolongation of QT/QTc interval (repeated exhibition of a QTc interval > 480 ms for both male and female patients)
14. No history of additional risk factors for torsade de pointes (e.g. clinically significant heart failure, hypokalemia, immediate family history of Long QT Syndrome)
15. Allow only patients who experienced relapse after 1 year from previous HiDAC treatment or who didn't receive HiDAC previously (Note: This inclusion applies only to South Korea)

EXCLUSION CRITERIA:

1. Patients who have received cytotoxic chemotherapy treatment for their current relapsed or refractory AML. (Treatment with hypomethylating agents (decitabine or azacytidine) either alone or in combination with venetoclax are allowed until the day prior to starting of CHAM or HAM therapy and control sub-groups (MEC and FLAG). Targeted therapies including FLT3 or IDH1/2 inhibitors and/or Hydrea and/or venetoclax are allowed. Targeted therapies and Hydrea may be taken until the day prior to starting CHAM or HAM therapy or control sub-groups (MEC and FLAG)
2. Vulnerable adult and patient whose health conditions does not allow them to give their consent
3. History or evidence of any other clinically significant disorder, condition or disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, symptomatic myocardial infection, uncontrolled cardiac arrhythmia, pericardial disease or heart failure New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity and in the opinion of the Investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures or completion
4. Patients with active Central Nervous System (CNS) involvement (leukemic infiltration, blast in the spinal fluid)
5. Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g. active peptic ulcer disease)
6. Female patients who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 months after the last dose of CHAM or HAM therapy or control sub-groups, MEC and FLAG (the teratogenic potential of CPI-613® (devimistat) is unknown). Female patients of childbearing potential with a positive pregnancy test assessed by a serum pregnancy test at Screening
7. Women of childbearing potential (i.e. women who are pre-menopausal or < 2 years postmenopausal or not surgically sterile) unwilling to practice a highly effective method of birth control consistent with local regulations regarding the use of birth control methods during treatment and for 6 months after completion of CHAM or HAM therapy or control sub-groups, MEC and FLAG for AML
8. Male patients with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for 6 months after completion of CHAM or HAM therapy or control sub-groups, MEC and FLAG
9. Male patients unwilling to abstain from donating sperm during treatment and for 6 months after completion of CHAM or HAM therapy or control sub-groups, MEC and FLAG with potential highest teratogenic risk
10. Known hypersensitivity to study treatment drugs or any of the excipient(s) contained in the drug formulation
11. Life expectancy less than 3 months
12. Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
13. Unwilling or unable to follow protocol requirements
14. Patients with large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly)
15. Patients with any amount of clinically significant pericardial effusion that requires drainage.
16. Evidence of ongoing, uncontrolled bacterial, viral or fungal infection
17. Patients with known human immunodeficiency virus infection
18. History of other malignancy within the past 5 years, with the following exception(s):

    1. Malignancy treated with curative intent and with no known active disease present for ≥ 5 years before enrolment and felt to be at low risk for recurrence by the treating physician
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of recurrent or residual disease
    3. Adequately treated cervical carcinoma in situ without evidence of disease
    4. Prostate cancer Stage 1
19. Patients receiving any other standard or investigational treatment for AML, or any other investigational agent for any indication within the past 1 week prior to initiation of CPI-613® (devimistat) treatment (the use of Hydrea and/or venetoclax, oral tyrosine kinase inhibitors FLT3 or IDH 1/2 inhibitors are allowed until the day prior to starting CHAM or HAM therapy or control sub-groups, MEC and FLAG. Previous exposure to a hypomethylating agent either alone or in combination with venetoclax are allowed until the day prior to starting of CHAM or HAM therapy and control sub-groups (MEC and FLAG))
20. Patients who have received immunotherapy of any type within the past 1 week prior to initiation of CPI-613® (devimistat) treatment
21. Requirement for immediate palliative treatment of any kind including minor surgery
22. Patients who have received a chemotherapy regimen with autologous stem cell support (bone marrow transplantation) within 6 months of starting CHAM or HAM therapy or control sub-groups (MEC and FLAG)
23. Patients who have had allogenic bone marrow transplantation within the last 6 months. Patients who have had an allogenic transplant more than 6 months ago are eligible provided they have no graft vs host disease. (Note: Exclude only patients with active GVHD requiring therapy with immunosuppressive agents and not patients with stable GVHD not requiring immunosuppression.)
24. Cytarabine contraindications

    * Hypersensitivity to the cytarabine or to any of the excipients of cytarabine injection
    * Anemia, leucopenia and thrombocytopenia of non-malignant aetiology (e.g bone marrow aplasia); unless the clinician feels that such management offers the most hopeful alternative for the patient
    * Degenerative and toxic encephalopathies, especially after the use of methotrexate or treatment with ionizing radiation
25. Mitoxantrone contraindications

    * Mitoxantrone Sterile Concentrate is contraindicated in patients who have demonstrated prior hypersensitivity to mitoxantrone hydrochloride, other anthracyclines or any of its components. Use in patients with profound bone marrow suppression is a relative contraindication depending on the clinical circumstances
    * Mitoxantrone Sterile Concentrate should not be used during pregnancy or lactation
26. Strong CYP450 inducers should be prohibited
27. Etoposide contraindications

    •. Contraindicated in patients with a history of a severe hypersensitivity reaction to etoposide products
28. Fludarabine contraindications

    •. Contraindicated in those patients who are hypersensitive to this drug or its components
29. Filgrastim contraindications •. Contraindicated in patients with known hypersensitivity to E coli-derived proteins, Filgrastim, or any component of the product

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — Augusta University
Locations (60):
- United States (23):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Chao Family Comprehensive Cancer Center (University of California Irvine), Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa-Holden Cancer Care Center, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Atlantic Health System, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Stony Brook University Hospital, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - MD Andrson Cancer Center, Houston, Texas
  - Baylor Temple (BSW), Temple, Texas
  - University of Virginia, Charlottesville, Virginia
- Australia (4):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - Universitätsklinik für Innere Medizin, Graz
  - Paracelsus Medical University, Salzburg
  - Hanuschkrankenhaus der WGKK, Vienna
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Clinique Universitaire St Luc, Brussels
  - UN Gent, Ghent
- France (9):
  - Centre Hospitalier de Versailles - Hôpital André Mignot, Le Chesnay, Yvelines
  - CHU Amiens, Amiens
  - Service d'Hématologie Clinique, Hôpital Avicenne-APHP-Université Paris, Bobigny
  - CHU de Caen, Caen
  - Centre Hospitalier Universitaire Grenoble Hopital Michalon, Grenoble
  - CHU la Conecption, Marseille
  - CHU de Nice, Nice
  - Hopital Saint Louis, Paris
  - Centre hospitalier Lyon Sud, Pierre-Bénite
- Germany (4):
  - Klinikum Frankfurt Hoechst, Frankfurt
  - UniversitatsklinikumUKSH Kiel, Kiel
  - Universitatsklinikum Marburg, Marburg
  - Robert-Bosch- Krankenhaus, Stuttgart
- Poland (3):
  - Zespół Szpitali Miejskich w Chorzowie, Chorzów
  - Uniwersyteckie Centrum Kliniczne Klinika Hematologii i Transplantologii, Gdansk
  - Katedra i Klinika Hematologii, Wroclaw
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Institut Catala d'Oncologia (ICO) - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Son ESPASES, Palma de Mallorca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital U. P. La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pardee TS, Powell BL, Larson RA, Maly J, Keng M, Foster M, Choi EJ, Sill H, Cluzeau T, Jeyakumar D, Frankfurt O, Patel P, Schuster M, Koller E, Costello R, Platzbecker U, Montesinos P, Vives S, Nazha A, Cook R, Vigil-Gonzales C, Chantepie S, Luther S, Cortes J. Devimistat plus chemotherapy vs chemotherapy alone for older relapsed or refractory patients with AML: results of the ARMADA trial. Blood Neoplasia. 2024 Mar 29;1(2):100009. doi: 10.1016/j.bneo.2024.100009. eCollection 2024 Jun. PMID 40454396

RESULTS

PARTICIPANT FLOW:
Groups:
- CPI-613 + HD Cytarabine and Mitoxantrone: CPI-613 at 2,000 mg/m2/day from day 1 to 5.
  Cytarabine at 1gm/m2 (5 doses), every 12 hours starting day 3. Mitoxantrone at 6gm/m2 (3 doses), everyday following the 1st, 2nd and 5th doses of Cytarabine.
- Control (HAM) and Control Sub-groups (MEC and FLAG): Cytarabine at 1gm/m2 (5 doses), every 12 hours starting day 3. Mitoxantrone at 6gm/m2 (3 doses), everyday following the 1st, 3rd and 5th doses of Cytarabine.
  Mitoxantrone, Etoposide and Cytarabine
  Etoposide 80mg/m over 60 minutes as a central line IV infusion; 6 doses Day 1 though 6 Cytarabine 1000mg/m2 over 3 hours as a central line IV infusion: 6 doses, Day 1 through 6 Mitoxantrone 6 mg/m2 over 30 minutes as a central line IV infusion: 6 dose, Day 1 through 6
  Fludarabine, Cytarabine and Filgrastim
  Fludarabine 30mg/m2/day over 30 minutes as a central line IV infusion; 5 doses Day 1 though 5 Cytarabine 2g/m2 over 4 hours as a central line IV infusion: 4 hours after Fludarabine: 5 doses, Day 1 through 5 Filgrastim 5µg/kg/day by SQ or as per institutional guidelines starting from Day 1 through Day 5
Period: Overall Study
Arm/Group | CPI-613 + HD Cytarabine and Mitoxantrone | Control (HAM) and Control Sub-groups (MEC and FLAG)
Started | 98 | 102
Completed | 11 | 11
Not Completed | 87 | 91

BASELINE CHARACTERISTICS:
Population: All subjects randomized were included in the analysis. Post interim analysis, the study was discontinued and no additional data was collected and analyzed.
Groups:
- CPI-613 + HD Cytarabine and Mitoxantrone: CPI-613 + High Dose Cytarabine and Mitoxantrone
  CPI-613 at 2,000 mg/m2/day from day 1 to 5.
  Cytarabine at 1gm/m2 (5 doses), every 12 hours starting day 3. Mitoxantrone at 6gm/m2 (3 doses), everyday following the 1st, 2nd and 5th doses of Cytarabine.
  CPI-613 + High Dose Cytarabine and Mitoxantrone: CPI-613 + High Dose Cytarabine and Mitoxantrone CPI-613: 2000mg/m2, 5 doses once a day, days 1-5 Cytarabine 1gm/m2, 5 doses every 12hrs starting day 3 through day 5 Mitoxantrone 6mg/m2, 3 doses, once a day following the first, third and fifth doses of Cytarabine
- Total: Total of all reporting groups
Arm/Group | CPI-613 + HD Cytarabine and Mitoxantrone | Control (HAM) and Control Sub-groups (MEC and FLAG) | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 46 | 88
  >=65 years | 56 | 56 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 79
  Male | 61 | 60 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 72 | 81 | 153
  Unknown or Not Reported | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR)
Description: Complete disappearance of all clinical evidence of disease
Time Frame: 12 months
Population: Number of Participants with Complete Remission (CR)
Measure: Count of Participants; unit: Participants
Arm/Group | CPI-613 + HD Cytarabine and Mitoxantrone | Control (HAM) and Control Sub-groups (MEC and FLAG)
Number analyzed (Participants) | 98 | 102
Participants | 20 | 22

ADVERSE EVENTS:
Time Frame: 38 months
Arm/Group | CPI-613 + HD Cytarabine and Mitoxantrone | Control (HAM) and Control Sub-groups (MEC and FLAG)
All-Cause Mortality (participants affected / at risk) | 52/96 | 55/97
Serious Adverse Events (participants affected / at risk) | 36/96 | 34/97
Other Adverse Events (participants affected / at risk) | 93/96 | 94/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPI-613 + HD Cytarabine and Mitoxantrone (N=96) | Control (HAM) and Control Sub-groups (MEC and FLAG) (N=97)
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 6
Hemolysis (Blood and lymphatic system disorders) | 2 | 0
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
cardiac failure acute (Cardiac disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Achromobacter infection (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 0
Bacillus bacteraemia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Covid-19 (Infections and infestations) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 5
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 5
Septic Shock (Infections and infestations) | 3 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
device occlusion (Product Issues) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPI-613 + HD Cytarabine and Mitoxantrone (N=96) | Control (HAM) and Control Sub-groups (MEC and FLAG) (N=97)
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Achromobacter infection (Infections and infestations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Ageusia (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 9 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 35
Anal fistula (Gastrointestinal disorders) | 2 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 6
Aspergilloma (Infections and infestations) | 1 | 9
Aspergillus infection (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 3 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Atrial fibrillation (Cardiac disorders) | 7 | 1
Atrial flutter (Cardiac disorders) | 1 | 4
Atrioventricular block first degree (Cardiac disorders) | 1 | 1
Bacillus bacteraemia (Infections and infestations) | 1 | 0
Bacillus infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Bacteraemia (Infections and infestations) | 3 | 8
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 7
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 10 | 1
Blood creatinine increased (Investigations) | 2 | 5
Blood fibrinogen decreased (Investigations) | 0 | 7
Blood fibrinogen increased (Investigations) | 1 | 6
Blood folate decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood phosphorus increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 0 | 2
Body temperature increased (Investigations) | 0 | 0
Bone abscess (Infections and infestations) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 4 | 0
Breath sounds abnormal (Investigations) | 0 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 2
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 5 | 1
Candida infection (Infections and infestations) | 3 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Catheter management (Surgical and medical procedures) | 0 | 3
Catheter site erythema (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter site induration (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 2
Cellulitis (Infections and infestations) | 5 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 4
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 5 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 10
Circulatory collapse (Vascular disorders) | 1 | 0
Citrobacter infection (Infections and infestations) | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 4 | 0
Clostridium difficile infection (Infections and infestations) | 4 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 6 | 0
Conjunctivitis (Infections and infestations) | 0 | 2
Constipation (Gastrointestinal disorders) | 21 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 20
COVID-19 (Infections and infestations) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 9
Creatinine renal clearance decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 3
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Device related infection (Infections and infestations) | 3 | 0
Device related thrombosis (General disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 43 | 4
Disorientation (Psychiatric disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 22
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 8
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 3 | 2
Dyskinesia (Nervous system disorders) | 0 | 0
Dysmetria (Nervous system disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dysuria (Renal and urinary disorders) | 3 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 12
Ecthyma (Infections and infestations) | 1 | 1
Ejection fraction decreased (Investigations) | 3 | 3
Electrocardiogram abnormal (Investigations) | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 2
Endocarditis (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 12
Eye haemorrhage (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 1
Eye pruritus (Eye disorders) | 1 | 1
Eye swelling (Eye disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Fatigue (General disorders) | 15 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 35 | 2
Fibrin D dimer increased (Investigations) | 2 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 13
Flatulence (Gastrointestinal disorders) | 3 | 32
Fluid overload (Metabolism and nutrition disorders) | 4 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 5
Folliculitis (Infections and infestations) | 1 | 6
Fungal oesophagitis (Infections and infestations) | 0 | 0
Gait disturbance (General disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Generalised oedema (General disorders) | 2 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Gingival erythema (Gastrointestinal disorders) | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 1
Gingivitis (Infections and infestations) | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Graft versus host disease in skin (Immune system disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 6 | 0
Haemolysis (Blood and lymphatic system disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 0
Hallucination (Psychiatric disorders) | 2 | 2
Hallucination, visual (Psychiatric disorders) | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 3
Headache (Nervous system disorders) | 19 | 0
Heart rate increased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 23
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatosplenic candidiasis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkinesia (Nervous system disorders) | 0 | 10
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 | 1
Hypersensitivity (Immune system disorders) | 1 | 2
Hypertension (Vascular disorders) | 5 | 0
Hypertensive crisis (Vascular disorders) | 1 | 8
Hyperthermia (General disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 10
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 36
Hypophosphataemia (Metabolism and nutrition disorders) | 15 | 15
Hypotension (Vascular disorders) | 10 | 4
Hypothermia (General disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 14
Ileus (Gastrointestinal disorders) | 1 | 14
Infection (Infections and infestations) | 3 | 0
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Injection site reaction (General disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 10 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 2
Jugular vein thrombosis (Vascular disorders) | 1 | 8
Klebsiella bacteraemia (Infections and infestations) | 2 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 2
Leptotrichia infection (Infections and infestations) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0
Leuconostoc infection (Infections and infestations) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 0
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 4
Localised oedema (General disorders) | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 12 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 11
Medical device site pain (General disorders) | 2 | 0
Medical device site pruritus (General disorders) | 1 | 1
Mesenteric panniculitis (Gastrointestinal disorders) | 1 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0
Moraxella infection (Infections and infestations) | 0 | 0
Morganella infection (Infections and infestations) | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal herpes (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 31 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 25
Neutropenic colitis (Gastrointestinal disorders) | 1 | 2
Neutropenic sepsis (Infections and infestations) | 1 | 0
Neutrophil count decreased (Investigations) | 12 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Ocular discomfort (Eye disorders) | 1 | 15
Ocular hyperaemia (Eye disorders) | 1 | 1
Oedema peripheral (General disorders) | 19 | 1
Oral candidiasis (Infections and infestations) | 1 | 3
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1
Oral infection (Infections and infestations) | 2 | 20
Oral pain (Gastrointestinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Orthostatic hypotension (Vascular disorders) | 2 | 0
Pain (General disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 4
Pathogen resistance (Infections and infestations) | 0 | 5
Pericardial effusion (Cardiac disorders) | 2 | 2
Peripheral swelling (General disorders) | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Platelet count decreased (Investigations) | 19 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 20
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonia fungal (Infections and infestations) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 10
Polyneuropathy (Nervous system disorders) | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 5
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Prophylaxis of nausea and vomiting (Surgical and medical procedures) | 1 | 1
Prothrombin time prolonged (Investigations) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1
Pseudomonal bacteraemia (Infections and infestations) | 2 | 4
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonal skin infection (Infections and infestations) | 0 | 1
Psychogenic seizure (Nervous system disorders) | 0 | 4
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulse abnormal (Investigations) | 1 | 1
Pyrexia (General disorders) | 22 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 22
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 4
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 9
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 2
Rash pustular (Infections and infestations) | 2 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 2
Root canal infection (Infections and infestations) | 1 | 1
Scrotal infection (Infections and infestations) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Sepsis (Infections and infestations) | 10 | 1
Septic shock (Infections and infestations) | 5 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 10
Sinusitis (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin wound (Injury, poisoning and procedural complications) | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 3 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Stenotrophomonas sepsis (Infections and infestations) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 10 | 2
Stomatococcal infection (Infections and infestations) | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 2 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 15
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0
Swelling face (General disorders) | 0 | 0
Swelling of eyelid (Eye disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Taste disorder (Nervous system disorders) | 0 | 0
Terminal ileitis (Gastrointestinal disorders) | 1 | 2
Thirst (General disorders) | 0 | 4
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 14
Tooth infection (Infections and infestations) | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Transaminases increased (Investigations) | 2 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Troponin I increased (Investigations) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 1 | 2
Urinary hesitation (Renal and urinary disorders) | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 6
Urinary retention (Renal and urinary disorders) | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Vision blurred (Eye disorders) | 2 | 3
Visual acuity reduced (Eye disorders) | 1 | 0
Visual field defect (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 10 | 1
Vomiting projectile (Gastrointestinal disorders) | 0 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
White blood cell count decreased (Investigations) | 15 | 14
Wound (Injury, poisoning and procedural complications) | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 33 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Device occlusion (Product Issues) | 0 | 13
Vertigo positional (Ear and labyrinth disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03504410/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT03504410/SAP_001.pdf